CLINICAL TRIAL: NCT02329301
Title: Assessing the Effectiveness of Mass Drug Administration (MDA) With Dihydroartemisinin + Piperaquine for Reducing Malaria Parasite Infection Prevalence and Incidence in Southern Province Zambia
Brief Title: Mass Drug Administration With Dihydroartemisinin + Piperaquine for Reducing Malaria in Southern Zambia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PATH (Other)
Collaborators: Ministry of Health, Zambia (Other Government); Minister of Community Development, Mother and Child Health, Zambia (Other); Tulane University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PATH-WIRB-20140824
Record Dates: First submitted 2014-11-13; First posted 2014-12-31 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Malaria; Malaria, Falciparum
Keywords: malaria; malaria, falciparum; antimalarials
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Mass Drug Administration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MDA with DHAp (Eurartesim) (Experimental): All consenting community members eligible to receive DHAp will be provided age-appropriate treatment dose of DHAp regardless of the malaria rapid diagnostic test (RDT) result. Treatment will be administered in a house-to-house campaign.
  Interventions: Drug: MDA with DHAp (Eurartesim)
- Focal MDA with DHAp (Eurartesim) (Experimental): All consenting household members eligible to receive DHAp and living in a household where anyone in the household tests positive with a malaria rapid diagnostic test (RDT) will receive the age-appropriate treatment dose of DHAp. If no one in the household tests RDT positive then no one in the household will receive DHAp. Treatment will be administered in a house-to-house campaign.
  Interventions: Drug: Focal MDA with DHAp (Eurartesim)
- Standard of Care (Control) (No Intervention): The standard of care arm will reflect no community-based treatment interventions but will have the standard of care offered by the Ministry of Health and Ministry of Community Development, Mother and Child Health which applies to all arms. This includes available mosquito net coverage, indoor residual spraying and passive case detection of individuals seeking treatment from a health provider at a clinic or health post.

INTERVENTIONS:
Drug: MDA with DHAp (Eurartesim) — Eurartesim is the brand name.
  Other Names: mass drug administration with DHAp
  Arms: MDA with DHAp (Eurartesim)
Drug: Focal MDA with DHAp (Eurartesim) — Eurartesim is the brand name.
  Other Names: focal mass drug administration with DHAp
  Arms: Focal MDA with DHAp (Eurartesim)

SUMMARY:
To quantify the relative effectiveness, cost, and cost-effectiveness of fMDA and MDA with DHAp against no mass treatment for reducing P. falciparum parasite prevalence, confirmed OPD malaria case incidence and cohort infection incidence in areas of high and low malaria transmission and in a program-relevant manner that will permit adoption and adaptation for wider-scale deployment.

DETAILED DESCRIPTION:
To quantify the relative effectiveness, cost, and cost-effectiveness of fMDA and MDA with DHAp against no mass treatment for reducing P. falciparum parasite prevalence, confirmed OPD malaria case incidence and cohort infection incidence in areas of high and low malaria transmission and in a program-relevant manner that will permit adoption and adaptation for wider-scale deployment.

In areas stratified by high and low malaria transmission, are 2 rounds of fMDA and MDA with DHAp more effective than no mass treatment (current standard of care) at reducing malaria parasite prevalence, health facility confirmed case incidence and community infection incidence over a 12 month period

* Null hypothesis (H0): There is no benefit of 2 rounds of fMDA or MDA with DHAp over current standard of care (national policy of case management) at reducing malaria parasite prevalence, health facility confirmed case incidence and community infection incidence over a 12 month period.
* Research hypothesis (HR): 2 rounds of fMDA and MDA with DHAp during the low transmission season will be significantly more effective than no mass treatment (standard of care) at reducing malaria parasite prevalence, health facility confirmed case incidence and community infection incidence over a 12 month period.

The research objectives are:

1. In areas stratified by high and low malaria transmission, evaluate the relative effectiveness of 2 rounds of fMDA with DHAp (fMDA arm), 2 rounds of community-wide MDA with DHAp (MDA arm) and no mass treatment (current standard of care - control arm) on the outcomes of reducing malaria parasite prevalence, confirmed case incidence and infection incidence over a 12 month period;
2. In areas stratified by high and low malaria transmission, assess the percent of health facility catchment areas (HFCA) with fMDA and MDA interventions that are able to reduce annual confirmed malaria case incidence to below 25 cases per 1,000 catchment population, which would permit the transition to a passive case investigation approach for malaria elimination;
3. Quantify the population coverage of the fMDA and MDA interventions in the study areas, including the identification of systematic barriers to achieving high coverage, under best programmatic efforts using directly observed treatment (DOT) to assure full treatment;
4. Assess and compare the cost and cost-effectiveness of fMDA and MDA with DHAp to no mass treatment in areas of high and low transmission;
5. Assess the adherence of taking a full course of DHAp by the fMDA and MDA interventions in areas of high and low transmission, under best programmatic efforts using DOT to assure full treatment;
6. Assess the clearance of asexual stage parasites at day 7 following the administration of DHAp under the best programmatic efforts using DOT to assure full treatment; and
7. Assess the acceptability of participating in the fMDA and MDA interventions among community members and health care leaders in areas of high and low transmission.

The study population includes:

Population of ~560,000 people in ~112,000 households in 60 health facility catchment areas near Lake Kariba in Southern Province.

Cluster randomized controlled trial in high and low transmission areas will be used to evaluate the fMDA and MDA interventions against current standard of care for the effect on population-wide parasite prevalence (RDT and more sensitive assay), community cohort infection incidence and routinely collected confirmed malaria case incidence.

The primary outcomes are:

1. Parasite prevalence during the high transmission season among children <6 years old (excluding neonates <1 month)
2. Pf infection incidence rate among individuals ≥3 months
3. Total and confirmed outpatient (OPD) malaria case incidence and inpatient (IPD) malaria case incidence among all ages
4. RDT test positivity rate from fMDA and MDA interventions (plus control group)
5. Population coverage of the fMDA and MDA interventions at each round

The entire population will be included in the study; interventions will be grouped/assigned randomly according to health facility catchment area (n= 60 health facilities), matched on potential confounding factors. Household surveys in the high transmission season before and after the interventions will be used for ascertaining malaria parasite prevalence. A longitudinal cohort will be used for ascertaining the infection incidence rate. The health system rapid reporting system will be used for ascertaining confirmed malaria case incidence.

ELIGIBILITY:
Inclusion Criteria:

* anyone not excluded and consenting

Exclusion Criteria:

* contraindications from manufacturer for medications including currently taking haloperidol, artane, Phenergan (Promethazine), chlorpromazine, erythromycin, Azithromycin, clarithromycin, Ketoconazole, fluconazole, mefloquine (as prophylaxis), lumefantrine (in Coartem), quinine, Septrin
* anyone seriously ill
* currently taking antimalarial medicines
* allergy to artemisinin drugs
* pregnant women in first trimester
* children under 3 months of age
* reported heart condition

Min Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2430 (Actual)
Dates: Start 2014-09; Primary Completion 2016-06 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Parasite prevalence during the high transmission season among children <6 years old (excluding neonates <1 month) | For up to 12 months
  Parasite prevalence during the high transmission season among children <6 years old (excluding neonates <1 month)
P.falciparum infection incidence rate among individuals ≥3 months | For up to 12 months
  P.falciparum infection incidence rate among individuals ≥3 months

SECONDARY OUTCOMES:
Total and confirmed outpatient (OPD) malaria case incidence and inpatient (IPD) malaria case incidence among all ages | For up to 48 months (including retrospectively)
  Total and confirmed outpatient (OPD) malaria case incidence and inpatient (IPD) malaria case incidence among all ages
Malaria rapid diagnostic test test positivity rate from focal mass drug administration (fMDA) and mass drug administration (MDA) interventions (plus control group) | For up to 10 months
  Malaria rapid diagnostic test test positivity rate from focal mass drug administration (fMDA) and mass drug administration (MDA) interventions (plus control group)

OTHER OUTCOMES:
Population coverage of the fMDA and MDA interventions at each round | For up to 4 months
  Population coverage of the fMDA and MDA interventions at each round

CONTACTS AND LOCATIONS:
Overall Officials: John M Miller, PhD, Principal Investigator — PATH
Locations (1):
- Southern province medical office, Choma, Southern Province, Zambia

REFERENCES:
- [Background] Eisele TP, Silumbe K, Finn T, Chalwe V, Kamuliwo M, Hamainza B, Moonga H, Bennett A, Yukich J, Keating J, Steketee RW, Miller JM. Assessing the effectiveness of household-level focal mass drug administration and community-wide mass drug administration for reducing malaria parasite infection prevalence and incidence in Southern Province, Zambia: study protocol for a community randomized controlled trial. Trials. 2015 Aug 13;16:347. doi: 10.1186/s13063-015-0862-3. PMID 26268804
- [Background] Eisele TP, Bennett A, Silumbe K, Finn TP, Chalwe V, Kamuliwo M, Hamainza B, Moonga H, Kooma E, Chizema Kawesha E, Yukich J, Keating J, Porter T, Conner RO, Earle D, Steketee RW, Miller JM. Short-term Impact of Mass Drug Administration With Dihydroartemisinin Plus Piperaquine on Malaria in Southern Province Zambia: A Cluster-Randomized Controlled Trial. J Infect Dis. 2016 Dec 15;214(12):1831-1839. doi: 10.1093/infdis/jiw416. PMID 27923947
- [Background] Alonso PL. The Role of Mass Drug Administration of Antimalarials. Am J Trop Med Hyg. 2020 Aug;103(2_Suppl):1-2. doi: 10.4269/ajtmh.20-0729. No abstract available. PMID 32618264
- [Background] Eisele TP, Bennett A, Silumbe K, Finn TP, Porter TR, Chalwe V, Hamainza B, Moonga H, Kooma E, Chizema Kawesha E, Kamuliwo M, Yukich JO, Keating J, Schneider K, Conner RO, Earle D, Slutsker L, Steketee RW, Miller JM. Impact of Four Rounds of Mass Drug Administration with Dihydroartemisinin-Piperaquine Implemented in Southern Province, Zambia. Am J Trop Med Hyg. 2020 Aug;103(2_Suppl):7-18. doi: 10.4269/ajtmh.19-0659. PMID 32618247
- [Background] Yukich JO, Scott C, Silumbe K, Larson BA, Bennett A, Finn TP, Hamainza B, Conner RO, Porter TR, Keating J, Steketee RW, Eisele TP, Miller JM. Cost-Effectiveness of Focal Mass Drug Administration and Mass Drug Administration with Dihydroartemisinin-Piperaquine for Malaria Prevention in Southern Province, Zambia: Results of a Community-Randomized Controlled Trial. Am J Trop Med Hyg. 2020 Aug;103(2_Suppl):46-53. doi: 10.4269/ajtmh.19-0661. PMID 32618249
- [Background] Finn TP, Porter TR, Moonga H, Silumbe K, Daniels RF, Volkman SK, Yukich JO, Keating J, Bennett A, Steketee RW, Miller JM, Eisele TP. Adherence to Mass Drug Administration with Dihydroartemisinin-Piperaquine and Plasmodium falciparum Clearance in Southern Province, Zambia. Am J Trop Med Hyg. 2020 Aug;103(2_Suppl):37-45. doi: 10.4269/ajtmh.19-0667. PMID 32618267
- [Background] Finn TP, Yukich JO, Bennett A, Porter TR, Lungu C, Hamainza B, Chizema Kawesha E, Conner RO, Silumbe K, Steketee RW, Miller JM, Keating J, Eisele TP. Treatment Coverage Estimation for Mass Drug Administration for Malaria with Dihydroartemisinin-Piperaquine in Southern Province, Zambia. Am J Trop Med Hyg. 2020 Aug;103(2_Suppl):19-27. doi: 10.4269/ajtmh.19-0665. PMID 32618251
- [Background] Silumbe K, Finn TP, Jennings T, Sikombe C, Chiyende E, Hamainza B, Chizema Kawesha E, Eisele TP, Earle D, Steketee RW, Miller JM. Assessment of the Acceptability of Testing and Treatment during a Mass Drug Administration Trial for Malaria in Zambia Using Mixed Methods. Am J Trop Med Hyg. 2020 Aug;103(2_Suppl):28-36. doi: 10.4269/ajtmh.19-0663. PMID 32618242
- [Background] Miller JM, Eisele TP, Fraser MS, Lewis MT, Slutsker L, Chizema Kawesha E. Moving from Malaria Burden Reduction toward Elimination: An Evaluation of Mass Drug Administration in Southern Province, Zambia. Am J Trop Med Hyg. 2020 Aug;103(2_Suppl):3-6. doi: 10.4269/ajtmh.19-0669. PMID 32618265
- [Background] Bennett A, Porter TR, Mwenda MC, Yukich JO, Finn TP, Lungu C, Silumbe K, Mambwe B, Chishimba S, Mulube C, Bridges DJ, Hamainza B, Slutsker L, Steketee RW, Miller JM, Eisele TP. A Longitudinal Cohort to Monitor Malaria Infection Incidence during Mass Drug Administration in Southern Province, Zambia. Am J Trop Med Hyg. 2020 Aug;103(2_Suppl):54-65. doi: 10.4269/ajtmh.19-0657. PMID 32618245
- [Background] Chishimba S, Mwenda M, Mambwe B, Mulube C, Chalwe V, Moonga H, Hamainza B, Chizema-Kawesha E, Steketee RW, Domingo G, Fraser M, Kahn M, Pal S, Silumbe K, Conner RO, Bennett A, Porter TR, Eisele TP, Miller JM, Bridges DJ. Prevalence of Plasmodium falciparum and Non-falciparum Infections by Photo-Induced Electron Transfer-PCR in a Longitudinal Cohort of Individuals Enrolled in a Mass Drug Administration Trial in Southern Province, Zambia. Am J Trop Med Hyg. 2020 Aug;103(2_Suppl):82-89. doi: 10.4269/ajtmh.19-0668. PMID 32618252
- [Derived] Shah MP, Hwang J, Choi L, Lindblade KA, Kachur SP, Desai M. Mass drug administration for malaria. Cochrane Database Syst Rev. 2021 Sep 29;9(9):CD008846. doi: 10.1002/14651858.CD008846.pub3. PMID 34585740